CLINICAL TRIAL: NCT05201469
Title: A Phase 2a Randomized Placebo-Controlled Double-Blind Multicenter Trial of VIB4920 for Active Lupus Nephritis (ITN091AI)
Brief Title: VIBRANT: VIB4920 for Active Lupus Nephritis
Acronym: VIBRANT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DAIT ITN091AI
Record Dates: First submitted 2022-01-07; First posted 2022-01-21 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis; Mycophenolate mofetil; VIB4920
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VIB4920 (Experimental): Participants will receive VIB4920 1500 mg intravenously at Weeks 0, 2, 4, 8, 12, 16, 20, and 24.
  Participants who previously received 1000 mg of methylprednisolone IV within 42 days of Visit 0 will not receive additional methylprednisolone IV on Day 0. Participants who previously received less than 1000 mg of methylprednisolone IV within 42 days of Visit 0 will receive an additional dose of methylprednisolone IV at Day 0, according to the following formula, where X is the intravenous dose previously received and Y is the intravenous dose administered on Day 0: 1000 mg - X = Y. Participants will begin MMF 2-3 g per day and prednisone 25 mg per day, tapered to 5 mg per day by Week 8. The prednisone dose may be tapered more rapidly and to a dose lower than 5 mg/d, at the discretion of the site investigator. Prednisone of no more than 5 mg/d will be continued until Week 60.
  Interventions: Drug: VIB4920
- VIB4920 Placebo (Placebo Comparator): Participants will receive VIB4920 placebo intravenously at Weeks 0, 2, 4, 8, 12, 16, 20, and 24.
  Participants who previously received 1000 mg of methylprednisolone IV within 42 days of Visit 0 will not receive additional methylprednisolone IV on Day 0. Participants who previously received less than 1000 mg of methylprednisolone IV within 42 days of Visit 0 will receive an additional dose of methylprednisolone IV at Day 0, according to the following formula, where X is the intravenous dose previously received and Y is the intravenous dose administered on Day 0: 1000 mg - X = Y. Participants will begin MMF 2-3 g per day and prednisone 25 mg per day, tapered to 5 mg per day by Week 8. The prednisone dose may be tapered more rapidly and to a dose lower than 5 mg/d, at the discretion of the site investigator. Prednisone of no more than 5 mg/d will be continued until Week 60.
  Interventions: Drug: Placebo for VIB4920

INTERVENTIONS:
Drug: VIB4920 — Participants will receive 1500 mg of VIB4920 at Weeks 0, 2, 4, 8, 12, 16, 20, and 24 while continuing on MMF and prednisone
  Arms: VIB4920
Drug: Placebo for VIB4920 — Participants will receive placebo for VIB4920 at Weeks 0, 2, 4, 8, 12, 16, 20, and 24 while continuing on MMF and prednisone
  Arms: VIB4920 Placebo

SUMMARY:
This is a multi-center double-blind placebo controlled clinical trial evaluating the efficacy of VIB4920 combined with mycophenolate mofetil (MMF) and prednisone in achieving a renal response in participants with active lupus nephritis (LN).

DETAILED DESCRIPTION:
Seventy-four eligible participants with active lupus nephritis (LN) will be randomized to receive VIB4920 1500 mg or placebo intravenously at Weeks 0, 2, 4, 8, 12, 16, 20, and 24. Participants will receive a total of 1000 mg of methylprednisolone according to either of the following schedules:

* 1000 mg methylprednisolone IV at Day 0, or
* 500 mg methylprednisolone IV at Day 0 and at Day 1.

Participants who previously received 1000 mg of methylprednisolone IV within 42 days of Visit 0 will not receive additional methylprednisolone IV on Day 0. Participants who previously received less than 1000 mg of methylprednisolone IV within 42 days of Visit 0 will receive an additional dose of methylprednisolone IV at Day 0, according to the following formula, where X is the intravenous dose previously received and Y is the intravenous dose administered on Day 0: 1000 mg - X = Y. Participants will also receive MMF 2-3 g per day and will receive prednisone 25 mg/d beginning on Day 0, or on the day after completion of methylprednisolone. Prednisone will be tapered to 5 mg/d by Week 8.

ELIGIBILITY:
Inclusion Criteria:

Individuals who meet all of the following criteria are eligible for enrollment as study participants:

1. Age 18 years or older.
2. Classification of Systemic Lupus Erythematosus (SLE) by any of the following criteria: the 1997 update of the 1982 American College of Rheumatology (ACR) criteria, the 2012 Systemic Lupus International Collaborating Clinics (SLICC) criteria, or the 2019 European League Against Rheumatism (EULAR)/ACR criteria.
3. UPCR ≥ 1.0 based on a 24-hour urine collection at Visit -1 or within 14 days prior to Visit -1.
4. Renal biopsy within 24 weeks prior to Visit -1 of ISN/RPS LN with both of the following:

   1. Class III, Class IV, or Class V in combination with Class III or IV, and
   2. Modified NIH Activity Index ≥ 1.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for enrollment as study participants:

1. Inability or unwillingness to give written informed consent or comply with study protocol.
2. Contraindication to treatment with MMF or mycophenolate sodium; or treatment with MMF or mycophenolate sodium is inappropriate in the opinion of the investigator.
3. Treatment with a biologic agent, except belimumab, or investigational agent within 90 days or 5 half-lives prior to Visit 0, whichever is longer.
4. Rituximab or other B cell depleting agent within 6 months prior to Visit 0.
5. Prior treatment with VIB4920.
6. Receipt of a live attenuated vaccine within 4 weeks prior to Visit 0.
7. Comorbidities requiring treatment with systemic corticosteroids, including those that have required 3 or more courses of systemic corticosteroids within 12 months prior to Visit 0.
8. Current malignancy or history of malignancy, except for adequately treated basal cell carcinoma, squamous cell carcinoma, or cervical carcinoma in situ > 12 months prior to Visit 0.
9. ESRD, defined as eGFR < 20 ml/min/1.73m2.
10. History of transplantation.
11. The following risks for thromboembolic events:

    1. Recent or recurrent deep venous thrombosis or arterial thromboembolism.
    2. Immobilization or major surgery within 12 weeks prior to Visit 0.
    3. History of congenital or inherited deficiency of antithrombin III, protein S, or protein C.
    4. History of anti-phospholipid syndrome, according to the 2006 Sapporo classification criteria.
12. History of a severe allergy or hypersensitivity reaction to any component of the VIB4920 formulation.
13. Any one of the following laboratory abnormalities:

    1. Peripheral B cell count < 5/μl.
    2. Neutropenia (absolute neutrophil count < 1000/mm3).
    3. Anemia (hemoglobin < 8 g/dL).
    4. Thrombocytopenia (platelets < 50,000/mm3).
    5. Aspartate aminiotransferase or alanine aminotransferase ≥ 2x upper limit of normal.
14. Evidence of current or prior tuberculosis infection, including any of the following:

    1. Positive QuantiFERON-TB Gold or TB Gold Plus test.
    2. Positive T-SPOT.TB test.
    3. Positive purified protein derivation (PPD) tuberculin test, defined as > 5mm induration.
15. Human immunodeficiency virus (HIV) infection.
16. Current or past hepatitis B (HBV) infection.
17. Current or past hepatitis C virus (HCV) infection, except adequately treated HCV with documented sustained virologic response.
18. Active bacterial, viral, fungal, or opportunistic infection.
19. History of significant, recurrent, or chronic infection that may pose additional risks from participating in the study, in the opinion of the investigator.
20. History of severe psychiatric condition that would interfere with the participant's ability to comply with the study protocol, in the opinion of the investigator.
21. Current substance abuse, or history of substance abuse within 12 months of Visit 0.
22. Lack of peripheral venous access.
23. Pregnancy.
24. Breastfeeding.
25. Unwillingness to use a medically acceptable form of contraception for the duration of the study if female of child-bearing potential or if male with a partner of childbearing potential.
26. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving a complete renal response at week 36 | Week 36
  Complete renal response is defined as all of the following:
  1. Urine protein-to-creatinine ratio (UPCR) <= 0.5, based on a 24-hour urine collection
  2. Estimated glomerular filtration rate (eGFR) >= 120 ml/min/1.73 m^2 or, if < 120 ml/min/1.73 m^2, then >= 80 percent of the eGFR at baseline
  3. Prednisone <= 5 mg/day from Week 8, according to the prednisone dosing restrictions

SECONDARY OUTCOMES:
Proportion of participants who achieve a complete renal response | Weeks 12, 24, 48, and 60
  Complete renal response is defined as all of the following:
  1. Urine protein-to-creatinine ratio (UPCR) <= 0.5, based on a 24-hour urine collection
  2. Estimated glomerular filtration rate (eGFR) >= 120 ml/min/1.73 m^2 or, if < 120 ml/min/1.73 m^2, then > 80 percent of the eGFR at Week 0
  3. Prednisone tapered to <= 5 mg/day by Week 8, and adherence to the prednisone dosing restrictions
Proportion of participants who achieve an overall renal response | Weeks 12, 24, 36, 48 and 60
  Overall renal response is defined as all of the following:
  1. >= 50 percent improvement in the urine protein-to-creatinine ratio (UPCR) compared to baseline, based on a 24-hour urine collection
  2. Estimated glomerular filtration rate (eGFR) >= 120 ml/min/1.73 m^2, or if < 120 ml/min/1.73 m^2, then > 80 percent of the eGFR at baseline, and
  3. Prednisone <= 5 mg/day from Week 8, according to the prednisone dosing restrictions
Proportion of participants who achieve a BLISS-LN primary efficacy renal response (PERR) | Weeks 12, 24, 36, 48, and 60
  BLISS-LN primary efficacy renal response (PERR) defined as all of the following:
  1. UPCR ≤ 0.7, and
  2. eGFR ≥ 60 ml/min/1.73m2, or if < 60 ml/min/1.73m2, then ≥ 80% of the eGFR at baseline, and
  3. no receipt of a prohibited immunosuppressive or immunomodulatory medication
Urine Protein-to-Creatinine Ratio (UPCR) | Weeks 12, 24, 36, 48, and 60
  Based on 24-hour urine collection
Anti-dsDNA antibodies | Weeks 12, 24, 36, 48, and 60
  The change in the proportion of participants who had a negative anti-dsDNA test will be summarized by arm, and will be analyzed using an exact conditional logistic regression model
Change in proportion of participants with lower C3 levels after treatment initiation | Weeks 12, 24, 36, 48, and 60
  The change in the proportion of participants who were hypocomplementemic for C3 and C4 after initiation of VIB4920 or placebo will be summarized by arm, and analyzed using an exact conditional logistic regression model
Change in proportion of participants with lower C4 levels after treatment initiation | Weeks 12, 24, 36, 48, and 60
  The change in the proportion of participants who were hypocomplementemic for C3 and C4 after initiation of VIB4920 or placebo will be summarized by arm, and analyzed using an exact conditional logistic regression model
Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) | Weeks 12, 24, 36, 48, and 60
  The change in SLEDAI-2K scores after initiation of VIB4920 or placebo will be summarized by arm, and analyzed using an analysis of covariance (ANCOVA) model
Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index for Systemic Lupus Erythematosus (SLICC/ACR-DI) | Weeks 24 and 60
  The change in SLICC/ACR-DI scores after initiation of VIB4920 or placebo will be summarized by arm, and analyzed using an ANCOVA model
Proportion of participants who experience treatment failures | Week 0 to Week 60
  Treatment failure is defined as any one of the following:
  1. Receipt of SLE rescue therapy
  2. End-stage renal disease (ESRD), defined as eGFR < 20 ml/min/1.73m2
  3. Worsening of proteinuria or eGFR from Week 24 onward, defined as either:
     1. confirmed ≥ 50% increase in the UPCR to a value ≥ 3.0 compared to Visit -1, or
     2. confirmed ≥ 30% increase in eGFR to a value of < 60, compared to Visit -1
Number of participants who experience at least one serious adverse event | Week 0 to Week 60
  The number of participants who experienced at least one SAE and the number of participants who experienced at least one AESI will be analyzed using a Fisher's exact test.
Number of participants who experience at least one adverse Events of Special Interest | Week 0 to Week 60
  Adverse Events of Special Interests include:
  1. Anaphylaxis
  2. Grade 3 or greater infusion reaction
  3. Grade 3 or greater hypersensitivity reaction
  4. Grade 3 or greater infection
  5. Thromboembolic event
Change in Serum IgM over study participation | Weeks 12, 24, 36, 48, and 60
  Serum IgM levels will be analyzed using a longitudinal mixed effects model with the test results at the time points as the dependent variable
Change in Serum IgG over study participation | Weeks 12, 24, 36, 48, and 60
  Serum IgG levels will be analyzed using a longitudinal mixed effects model with the test results at the time points as the dependent variable

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dall'Era, M.D., Study Chair — University of California San Francisco School of Medicine: Lupus Clinic and Rheumatology Clinical Research Center; Betty Diamond, M.D., Study Chair — Feinstein Institute for Medical Research: Center for Autoimmune and Musculoskeletal Diseases; David Wofsy, M.D., Study Chair — University of California San Francisco School of Medicine: Lupus Clinic and Rheumatology Clinical Research Center
Locations (17):
- United States (17):
  - University of California San Diego School of Medicine: Division of Rheumatology, Allergy and Immunology, La Jolla, California
  - UCLA Medical Center: Division of Rheumatology, Los Angeles, California
  - of California, Irvine School of Medicine Division of Rheumatology, Orange, California
  - University of California San Francisco School of Medicine: Lupus Clinic and Rheumatology Clinical Research Center, San Francisco, California
  - University of Colorado School of Medicine: Division of Rheumatology, Aurora, Colorado
  - Yale University School of Medicine: Section of Rheumatology, New Haven, Connecticut
  - University of Miami Miller School of Medicine: Nephrology & Hypertension Division, Miami, Florida
  - Emory University School of Medicine: Division of Rheumatology, Atlanta, Georgia
  - University of Chicago, Department of Medicine: Rheumatology, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine in St. Louis: Division of Nephrology, St Louis, Missouri
  - Feinstein Institute for Medical Research: Center for Autoimmune and Musculoskeletal Diseases, Manhasset, New York
  - Hospital for Special Surgery, New York: Division of Rheumatology, New York, New York
  - Columbia University Medical Center: Department of Medicine, Division of Rheumatology, New York, New York
  - Penn State Health Milton S. Hershey Medical Center: Division of Rheumatology, Hershey, Pennsylvania
  - Temple University, Lewis Katz School of Medicine, Department of Medicine: Nephrology, Philadelphia, Pennsylvania
  - University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: Yes
Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical mechanistic data from NIAID/DAIT-funded grants and contracts
Time Frame: Within 24 months after database lock for the trial
Access Criteria: Open Access
URL: http://www.immport.org/home

REFERENCES:
- See also: Immune Tolerance Network (ITN) — https://www.immunetolerance.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait